CLINICAL TRIAL: NCT05058131
Title: The Effects of Fermentable Dietary Fibre Supplementation on Intestinal Permeability and Inflammation in Microscopic Colitis
Brief Title: Modulation of Intestinal Barrier Function and Inflammation Via Butyrate-promoting Dietary Fibre
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Robert Brummer, Professor, Örebro University, Sweden
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: MC-DF
Record Dates: First submitted 2021-09-09; First posted 2021-09-27 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Microscopic Colitis
MeSH Terms: conditions — Colitis, Microscopic | interventions — Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary fibre (Active Comparator): Butyrate-promoting dietary fibre
  Interventions: Dietary Supplement: Dietary fibre
- Placebo compound (Placebo Comparator): Placebo compound
  Interventions: Dietary Supplement: Placebo compound

INTERVENTIONS:
Dietary Supplement: Dietary fibre — Dietary fibre as a powder, 24 g per day for 6 weeks
  Arms: Dietary fibre
Dietary Supplement: Placebo compound — Maltodextrin powder, 24 g per day for 6 weeks
  Arms: Placebo compound

SUMMARY:
This study examines how a fermentable dietary fibre known to promote butyrate production impacts intestinal barrier function, intestinal microbiota, intestinal inflammation, and gastrointestinal symptoms in patients with microscopic colitis.

DETAILED DESCRIPTION:
The study examines the effects of a 6-week supplementation period with a dietary fibre product (type of wheat bran) on intestinal barrier function, intestinal inflammation, intestinal microbiota, and gastrointestinal symptoms in patients with MC. The study subjects will consume the study products (placebo-fibre, butyrate-promoting fibre) as a powder supplemented to their daily habitual diet. A maltodextrin-based product is used as placebo. After giving their informed consent, the study subjects fill out a background questionnaire to assess their eligibility for the study (Visit 1). Participants deemed suitable for the study will be randomised into two study arms (placebo-fibre, butyrate-promoting fibre) before undergoing a baseline visit (Visit 2) before the start of the intervention period. After the 6-week intervention period, the participants will come back for a final visit (Visit 3). In vivo intestinal permeability will be measured using the standard multi-sugar test at visits 2 and 3. Blood and faecal samples will also be collected during visits 2 and 3. In addition to the visits described above, a subset of patients (max. 20) will undergo a colonoscopy before and at the end of the intervention period at Örebro University Hospital where an experienced gastroenterologist collects 16 colonic biopsies. These colonic biopsies are mounted in an Ussing chamber system to specifically study colonic permeability. During visits 2 and 3, the participants also complete questionnaires to assess their gastrointestinal symptoms, quality of life, physical activity, and dietary habits. During the study period, the participants will also keep a daily diary recording the number of diarrheal and loose stools. The participants are asked to maintain their habitual diet and lifestyle as well as not to consume probiotic or prebiotic supplements.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Diagnosis of microscopic colitis (collagenous or lymphocytic colitis)
3. Active disease with no medication (e.g. budesonide) or stable budesonide treatment with or without symptoms
4. Age between 18-75

Exclusion Criteria:

1. Previous diagnosis of other organic gastrointestinal disease that interferes with the outcome parameters used in this study (e.g. ulcerative colitis)
2. Previous abdominal surgery which might influence gastrointestinal function, except appendectomy and cholecystectomy
3. History of or present gastrointestinal malignancy or polyposis
4. Diagnosis of gastrointestinal infection within the last 6 months
5. Current diagnosis of dementia, severe depression, major psychiatric disorder, or other incapacity for adequate cooperation
6. Chronic neurological/neurodegenerative disease (e.g. Parkinson's disease)
7. Autoimmune disease (e.g. rheumatoid arthritis)
8. Chronic pain syndromes (e.g. fibromyalgia)
9. Chronic fatigue syndrome
10. Severe endometriosis
11. Coeliac disease
12. Diagnosis of lactose intolerance within the last 3 months
13. Pregnancy or breast-feeding
14. Regular intake of anti-inflammatory and/or other immunosuppressive medication than budesonide within the last 3 months
15. Intake of proton pump inhibitors (e.g. omeprazol) within the last 4 weeks
16. Use of anti-depressants within the last 3 months
17. Regular intake of mast cell stabilizing drugs (e.g. sodium cromoglycate) within the last 3 months
18. Antimicrobial treatment within the last 12 weeks before baseline sampling
19. Antimicrobial prophylaxis (e.g. urinary tract infection)
20. Regular intake of probiotics, nutritional supplements, or herb products that might affect intestinal function within the last 4 weeks if the investigator considers that those could affect study outcome
21. Inability to maintain current diet and lifestyle during the study period
22. Alcohol or drug abuse
23. Any clinically significant present or past disease/condition which the investigator considers to possibly interfere with the study outcome

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Colonic permeability in vivo | 6 weeks
  Difference in urinary sucralose/erythritol excretion ratio between the study arms

SECONDARY OUTCOMES:
Small intestinal permeability in vivo | 6 weeks
  Difference in urinary lactulose/rhamnose excretion ratio between the study arms
Colonic permeability ex vivo in Ussing chambers | 6 weeks
  Difference in the translocation of FITC-labeled dextran and horseradish peroxidase between the study arms
Concentrations of intestinal fatty-acid binding protein | 6 weeks
  Difference in plasma concentrations of intestinal fatty-acid binding protein between the study arms
Concentrations of lipopolysaccharide-binding protein | 6 weeks
  Difference in plasma levels of lipopolysaccharide-binding protein between the study arms
Concentratios of faecal calprotectin | 6 weeks
  Difference in faecal levels of calprotectin between the study arms
Concentrations of faecal myeloperoxidase | 6 weeks
  Difference in faecal levels of myeloperoxidase between the study arms
Concentrations of high-sensitive C-reactive protein | 6 weeks
  Difference in plasma levels of high-sensitive C-reactive protein between the study arms
Concentrations of inflammatory cytokines | 6 weeks
  Difference in TNF-a, IFN-y, IL-1B, IL-4, IL-6, IL-8, IL-10 levels in serum between the study arms
Composition of intestinal microbiota | 6 weeks
  Difference in the composition of intestinal microbiota between the study arms
Functionality of intestinal microbiota | 6 weeks
  Difference in the levels of intestinal microbiota -derived metabolites in the serum and faeces between the study arms

OTHER OUTCOMES:
Faecal output measured by a daily diary | 6 weeks
  Difference in the number of diarrhoeal stools per day between the study arms
Gastrointestinal symptoms measured by Gastrointestinal Symptom Rating Scale | 6 weeks
  Difference in the frequency and severity of gastrointestinal symptoms between the study arms (15 questions with a scale of 1-7, minimum value 1, maximum 7, higher score correspond to a worse outcome)
Quality of life measured by EQ-5D-5L questionnaire | 6 weeks
  Difference in the scores of the quality of life between the study arms (Visual Analog Scale 0-100, lower value corresponds to a worse outcome)
Anxiety and depression measured by Hospital Anxiety and Depression Scale | 6 weeks
  Difference in the scores of anxiety and depression between the study arms (depression and anxiety scores separately, 7 questions each with a scale of 0-3, minimum score 0, maximum score 21 in both, higher value corresponds to a worse outcome)
General well-being measured by Short Health Scale | 6 weeks
  Difference in the scores of general well-being between the study arms (4 questions with a scale of 1-7, higher scores correspond to a worse outcome)
Concentrations of systemic and faecal markers of oxidative stress | 6 weeks
  Difference in blood and faecal markers of oxidative stress (e.g. glutathione) between the study arms
Concentrations of faecal chromogranins | 6 weeks
  Difference in faecal levels of chromogranins between the study arms

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Brummer, MD, PhD, Principal Investigator — Örebro University, Sweden
Locations (1):
- Örebro University, Örebro, Örebro County, Sweden

IPD SHARING:
Plan to Share IPD: No